CLINICAL TRIAL: NCT00004776
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Oral Topiramate for Lennox-Gastaut Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of California, Los Angeles (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11821; UCLA-567
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Lennox-Gastaut Syndrome
Keywords: Lennox-Gastaut syndrome; epilepsy; neurologic and psychiatric disorders; rare disease; seizures
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epilepsy; Neurologic Manifestations; Mental Disorders; Rare Diseases; Seizures | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
OBJECTIVES:

I. Evaluate the safety and efficacy of oral topiramate in patients with Lennox-Gastaut syndrome.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Following a 28-day baseline period, patients are randomly assigned to oral topiramate or placebo. The dose of study medication is titrated over the first 3 weeks; the maintenance dose is administered for the next 5 weeks.

Extended topiramate treatment is available to all patients after randomized therapy.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Lennox-Gastaut syndrome Slow spike and wave pattern on electroencephalogram At least 60 seizures with atypical absence and drop attacks within 1 month Seizure types allowed in addition to those above: Tonic Tonic-clonic Myoclonic Minor motor Absence of progressive lesion confirmed by computerized tomography or magnetic resonance imaging No change documented by physical exam subsequent to imaging No generalized status epilepticus within 3 months while complying with drug therapy No seizures resulting from progressive disease, e.g.: Active infection Neoplasm Metabolic disorder No anoxic episode requiring resuscitation within 1 year --Prior/Concurrent Therapy--

1 or 2 concurrent maintenance antiepileptics required At least 6 months since corticotropin At least 60 days since acetazolamide or zonisamide At least 60 days since investigational drug or device No ketogenic diet --Patient Characteristics-- Hematopoietic: No hematological abnormality within 2 years Hepatic: No hepatic disease within 2 years Renal: No nephrolithiasis No other renal disease within 2 years Cardiovascular: No clinically significant electrocardiographic abnormality No cardiovascular disease within 2 years Pulmonary: No respiratory disease within 2 years Other: Weight at least 25 lb (11.5 kg) No medical disease within 2 years, e.g.: Rheumatic fever Gastrointestinal abnormality Malignancy No psychiatric or mood disorder inconsistent with Lennox-Gastaut within 6 months requiring any of the following: Electroconvulsive therapy Antidepressants Anxiolytics Antipsychotics Lithium carbonate No history of alcohol or drug abuse No history of poor compliance on past antiepileptic therapy Able to take medication and maintain seizure calendar (assistance allowed) Adequate parental supervision 1 parent/guardian with adequate English fluency if English not patient's primary language The following required of fertile women: Negative serum-beta pregnancy test immediately prior to entry Normal menstrual flow for 3 months prior to entry Medically acceptable form of contraception during study

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10
Dates: Start 1993-11

CONTACTS AND LOCATIONS:
Overall Officials: W. Donald Shields, Study Chair — University of California, Los Angeles